CLINICAL TRIAL: NCT04346667
Title: Use and Dosage of Hydroxychloroquine and Chloroquine to Convert Real Time Polymerase Chain Reaction (RT-PCR) Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Coronavirus Infectious Disease 2019 (COVID-19) Patients to RT- PCR-Negative as a Means to Reduce Hospitalization Rate
Brief Title: Post-Exposure Prophylaxis for Asymptomatic SARS-CoV-2 COVID-19 Patients With choloroquinE Compounds
Acronym: PEACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual.
Sponsor: Government of Punjab, Specialized Healthcare and Medical Education Department (Other Government)
Collaborators: Mayo Hospital Lahore (Other); Services Institute of Medical Sciences, Pakistan (Other Government); Pakistan Kidney and Liver Institute (Unknown); Forman Christian College, Pakistan (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ammar Sarwar, Assistant Professor of Radiology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBC-COVID19-02
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2; Coronavirus Infection; Asymptomatic Condition; COVID-19
MeSH Terms: conditions — Coronavirus Infections; Asymptomatic Diseases; COVID-19 | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Active Comparator): Hydroxychloroquine loading dose (400 mg BID for 2 days) followed by 200 mg BID for 4 days plus standard of care
  Interventions: Drug: Hydroxychloroquine Sulfate Regular dose
- Arm 2 (Experimental): Hydroxychloroquine loading dose (400 mg BID) alone plus standard of care
  Interventions: Drug: Hydroxychloroquine Sulfate Loading Dose
- Arm 3 (Active Comparator): Chloroquine 500 mg BID for 5 days plus standard of care
  Interventions: Drug: Chloroquine
- Arm 4 (Placebo Comparator): Standard of care plus placebo (cannot be treated with hydroxychloroquine or chloroquine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Regular dose — Hydroxychloroquine administered based off of in-vitro pharmacokinetics study of optimal dosage for efficacy against SARS-CoV-2
  Arms: Arm 1
Drug: Hydroxychloroquine Sulfate Loading Dose — Hydroxychloroquine administered as a loading dose only
  Arms: Arm 2
Drug: Chloroquine — Chloroquine administered based off of in-vitro pharmacokinetics study of optimal dosage for efficacy against SARS-CoV-2
  Arms: Arm 3
Drug: Placebo — Standard of Care plus placebo
  Arms: Arm 4

SUMMARY:
To create a protocol for treatment of Pakistani patients with SARS-CoV-2 infection with an intent to reduce burden on institutional healthcare services by determining efficacy of different quinone drug dosing regimens in controlling SARS-CoV-2 infection for asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Nasopharyngeal RT-PCR positive SARS-CoV-2 patient
2. Age 20-50 years
3. BMI 18-28 kg/m2
4. Informed consent

Exclusion Criteria:

1. Symptoms: Cough, fever, shortness of breath
2. O2 saturation by pulse-oximeter below 94%
3. Co-morbidities: any pre-existing cardiac disease, pulmonary disease, diabetes
4. Arrhythmias and/or history of arrythmia
5. Psoriasis and/or history of psoriasis
6. Neuropathy or myopathy and/or history of these
7. Hypoglycemia and/or history of hypoglycemia
8. Pre-existing hepatic disease
9. Pre-existing renal disease
10. Use of antacids within 1 week
11. Use of antibiotics within 1 week
12. Pregnancy
13. RT-PCR performed >3 days prior to enrollment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
RT-PCR negative status | 6-7 days
  Percentage of patients who become RT-PCR negative with two RT-PCR tests performed at day 6 and day 7

SECONDARY OUTCOMES:
Progression of symptoms | 7 days
  Time to progression to next stage of SARS-CoV-2 disease severity index
Development of Symptoms | 7 days
  Time to onset of fever (temperature greater than 100 degree F), cough, or shortness of breath (respiratory rate >22 per minute).
Adverse events | 7 days
  Drug related adverse events as determined by data safety and monitoring board (DSMB)

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Expo Covid Center, Lahore, Punjab Province
  - Mayo Hospital, Lahore, Punjab Province
  - Pakistan Kidney and Liver Institute, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No